CLINICAL TRIAL: NCT05041504
Title: A Web-based Peer Navigation Program for Men With Prostate Cancer: A Hybrid Effectiveness-Implementation Trial
Brief Title: A Web-based Peer Navigation Program for Men With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of British Columbia (Other); Dalhousie University (Other); University of Toronto (Other); Canadian Cancer Society (CCS) (Other); Canadian Partnership Against Cancer (Unknown); Movember Foundation (Other); Walnut Foundation (Unknown); Prostate Cancer Support - Toronto (Unknown); Prostate Cancer Group - Burnaby (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-5126; Peer Navigation pRCT (Other: UHN)
Record Dates: First submitted 2021-08-10; First posted 2021-09-13 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; navigation; peer support; web-based; patient activation
MeSH Terms: conditions — Prostatic Neoplasms; Patient Participation

STUDY DESIGN:
Intervention Model Description: This is a 2-arm pragmatic randomized controlled trial with an active wait-list control, and an embedded process evaluation. Participants in the intervention group will receive the True North Peer Navigation intervention. Participants in the active control group will receive access to an online health resource library and will be offered the True North Peer Navigation intervention after study completion.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants assigned to the intervention arm will receive the True North Peer Navigation intervention.
  Interventions: Behavioral: Peer navigation
- Active Waitlist Control (Other): Participants assigned to the control arm will receive usual care and access to an online health resource library. After completion of the study, they will receive the True North Peer Navigation intervention.
  Interventions: Other: Active wait list control

INTERVENTIONS:
Behavioral: Peer navigation — Participants in the intervention group will receive ongoing support from a trained peer navigator for 3 months after completing treatment for prostate cancer via the True North Peer Navigation website. Participants will be matched with a trained peer navigator who assesses needs and barriers to care, provides practical, informational, and emotional support, and empowers them to take a proactive role in their health. Participants will also have access to a health resource library on the True North Peer Navigation website that contains local and national resources about prostate cancer.
  Other Names: True North Peer Navigation
  Arms: Intervention
Other: Active wait list control — Participants in the active wait list control group will receive usual care and access to a health resource library on the True North Peer Navigation website that contains local and national resources about prostate cancer. After completion of the study, patients in the active wait list control group will be matched with a peer navigator.
  Other Names: Web-based educational wait list control
  Arms: Active Waitlist Control

SUMMARY:
One in nine Canadian men will be diagnosed with prostate cancer (PC) in their lifetime. Although all treatment options can be effective in controlling the disease, treatment side effects such as problems with erections and controlling the bladder can significantly affect men's quality of life. Many men with PC say they do not get relevant information and emotional support, and experience gaps in care when dealing with these difficult issues. Previous studies have shown that cancer patient navigation improves access to care and support, and reduces healthcare costs. The investigators developed True North Peer Navigation - a peer navigation program for men with PC and a peer navigator training course. Men are matched online with a trained peer navigator who provides practical information and emotional support through the cancer journey. A pilot evaluation showed that it is highly acceptable to patients and peer navigators, and improves patient quality of life, social support and ability to manage their health. In this study, the investigators will conduct a randomized controlled trial of the True North Peer Navigation program in cancer centres in Ontario, British Columbia and Nova Scotia. Patients will be randomly assigned to receive True North Peer Navigation or an active wait list control consisting of usual care with access to information on the True North Peer Navigation website. The investigators will evaluate the effect of the True North Peer Navigation program on patient outcomes such as their ability to take a more active role in their health, quality of life, social support and use of health care services. In addition, the investigators will evaluate how True North Peer Navigation was implemented, the experiences patients and peer navigators, the factors that make it easier or harder for people to deliver the program to patients in different settings, as well as the cost of delivering the program, which will help us learn how to spread the program across the country.

DETAILED DESCRIPTION:
Background: Prostate cancer (PC) is a highly prevalent condition affecting 1 in 9 Canadian men. While the 5-year survival rate for PC is 93%, treatment-related side effects, such as sexual dysfunction and urinary incontinence, can significantly affect quality of life. Men with PC lack access to relevant information and emotional support, and report gaps in supportive care when dealing with these difficult issues. Previous research has shown that cancer patient navigation improves the timeliness of care and support, and reduces healthcare costs. Engaging volunteer cancer survivors as navigators is less costly, provides peer support, and benefits the navigator by improving their psychosocial health. The investigators developed True North Peer Navigation - an evidence-based peer navigation program for men with PC and a competency-based peer navigator training course. Men are matched online with a trained peer navigator who assesses needs and barriers to care, provides practical, informational, and emotional support, and empowers them to take a proactive role in their health. A pilot study showed True North Peer Navigation is highly acceptable to patients and peer navigators, and associated with improvements in quality of life, social support and patient activation to manage health.

Aim: This project aims to advance knowledge on the effectiveness and implementation of a web-based peer navigation program for men after treatment for PC.

Specific Objectives:

1. To determine the effect of True North Peer Navigation on patient outcomes in men with PC; and
2. To evaluate the delivery of True North Peer Navigation in terms of fidelity, cost, and the experiences of patients and peer navigators, and to identify barriers and facilitators to its implementation in oncology settings.

Methods: Guided by the SPOR Patient Engagement Framework, the investigators will conduct a type-1 hybrid effectiveness-implementation study at cancer centres in Ontario, British Columbia and Nova Scotia. For objective 1, the investigators will conduct a pragmatic randomized controlled trial to evaluate the impact of True North Peer Navigation compared to an active wait list control on patient activation (primary) and needs, quality of life, anxiety, depression, fear of recurrence, social support, and access to services (secondary). One hundred and fifty-two patients (n=76 per arm) with PC will be recruited after treatment. Outcomes will be assessed at baseline (T0), 3-months (T1) and 6-months (T2). Objective 2 will involve a mixed-method process evaluation to investigate implementation fidelity, patient and navigator experiences, and cost-effectiveness of True North Peer Navigation, and to assess implementation barriers and facilitators with stakeholders informed by the Consolidated Framework for Implementation Research and the Theoretical Domains Framework.

Significance: True North Peer Navigation is an innovative solution to an important service gap in the lives of men with PC. This study has the potential to generate important evidence and strategies to support the implementation of peer navigation programs to improve the health outcomes of men with PC in Canada.

Note: The planned sample size described in the grant was 152 participants, considering an expected 35% dropout rate, and recruitment from three sites (PM, BC-Cancer and QEII). After the grant was awarded, we added two recruitment sites (VGH and Cape Breton Regional Hospital). As a result, the sample size was increased to 240 participants (also considering a 35% dropout rate) to address the expected increase in heterogeneity as recommended for pragmatic trials. However, recruitment at these sites was not possible due to insufficient clinical champion support. Hence, we reverted to our original planned sample size and ceased recruitment when it was reached.

ELIGIBILITY:
Inclusion Criteria:

1. Has been diagnosed with local, locally advanced or stable metastatic PC.
2. Has recently completed treatment within 3 months
3. Has an email address OR is willing to create one.
4. Can read and speak English.

Exclusion Criteria:

1. Has been diagnosed with advanced metastatic disease.
2. Is receiving palliative care.
3. Is not willing to be randomized.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Patient Activation at 3 months | 0, 3 months
  The primary outcome will be Patient Activation at 3 months. Patient Activation will be measured using the Patient Activation Measure (PAM). Higher scores represent a better outcome.

SECONDARY OUTCOMES:
Patient Activation at 6 months | 0, 6 months
  Patient Activation at 6 months will be assessed. Patient Activation will be measured using the Patient Activation Measure (PAM). Higher scores represent a better outcome.
Supportive Care Needs | 0, 3, 6 months
  Supportive Care Needs will be assessed at 3 months and 6 months separately. Supportive Care Needs will be measured with the 34-item Supportive Care Needs Survey-Short Form (SCNS-SF). Higher scores represent a worse outcome.
Health-Related Quality of Life | 0, 3, 6 months
  Health-related quality of life will be assessed at 3 months and 6 months separately. Health-related quality of life will be measured with the European Quality of Life, 5 Dimensions, 5 Levels (EQ-5D-5L) overall utility score. Higher scores represent a better outcome.
Prostate Cancer Quality of Life | 0, 3, 6 months
  Prostate Cancer Specific Quality of Life will be measured at 3 months and 6 months separately. Prostate Cancer Specific Quality of Life will be measured using the overall Patient-Oriented Prostate Utility Scale (PORPUS) score. Higher scores represent a better outcome.
Anxiety | 0, 3, 6 months
  Anxiety will be assessed at 3 months and 6 months separately. Anxiety will be measured using the Generalized Anxiety Disorder scale (GAD-7). Higher scores represent a worse outcome.
Depression | 0, 3, 6 months
  Depression will be assessed at 3 months and 6 months separately. Depression will be measured using the depression module of the Patient Health Questionnaire (PHQ-9). Higher scores represent a worse outcome.
Social Support | 0, 3, 6 months
  Social Support will be assessed at 3 months and 6 months separately. Social Support will be measured using the Enriched Social Support Scale, a multidimensional measure of perceived social support (ESSI). Higher scores represent a better outcome.
Fear of Cancer Recurrence | 0, 3, 6 months
  Fear of Cancer Recurrence will be assessed at 3 months and 6 months separately. Fear of Cancer Recurrence will be measured using the Fear of Cancer Recurrence Inventory -Short Form Scale (FCRI-SF). Higher scores represent a worse outcome.

OTHER OUTCOMES:
Quality-adjusted life year | 0,3,6 months
  An estimation of the combined health utility values derived from responses from the European Quality of Life, 5 Dimensions, 5 Levels (EQ-5D-5L) and length of life experienced by patient, between measurement time points.
Total healthcare costs | 3,6 months
  The total cost of publicly funded healthcare utilization (outside of delivery of the intervention) by patient while enrolled in the study. Number of times patient accessed publicly funded healthcare resources while enrolled in the study will be estimated based on the data gathered from the Health System Service Utilization Inventory (HSSUI). Resource use volumes will be used to micro-cost resource use costs such as physician care, allied health professional care, hospital care and pharmaceuticals.
Intervention cost | 3 years
  Incremental cost of the intervention (i.e., delivery of the peer navigation program not related to volunteer time, such as administrative costs, training costs, and overhead costs) will be estimated per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Bender, PhD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bender JL, Flora PK, Milosevic E, Soheilipour S, Maharaj N, Dirlea M, Parvin L, Matthew A, Kazanjian A. Training prostate cancer survivors and caregivers to be peer navigators: a blended online/in-person competency-based training program. Support Care Cancer. 2021 Mar;29(3):1235-1244. doi: 10.1007/s00520-020-05586-8. Epub 2020 Jul 2. PMID 32613373
- [Background] Flora PK, Bender JL, Miller AS, Parvin L, Soheilipour S, Maharaj N, Milosevic E, Matthew A, Kazanjian A. A core competency framework for prostate cancer peer navigation. Support Care Cancer. 2020 Jun;28(6):2605-2614. doi: 10.1007/s00520-019-05059-7. Epub 2019 Oct 15. PMID 31616997
- [Background] Maharaj N, Soheilipour S, Bender JL, Kazanjian A. Understanding Prostate Cancer Patients and Caregivers Support Needs: How Do They Manage Living with Cancer? Illness, Crisis & Loss. 2018; April 5:51-73.
- See also: TrueNORTH Peer Navigation intervention website — https://peernavigation.truenth.ca/start/pcc-i8/index.html